CLINICAL TRIAL: NCT02044913
Title: Randomized-controlled Trial of Aftercare-Coordination by Phone for Patients With Depression and Anxiety Subsequent to an Inpatient Treatment.
Brief Title: Randomized-controlled Trial of Aftercare-Coordination by Phone for Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0421-FSCP-Z202; 0421-FSCP-Z202 (Other Grant/Funding Number: 0421-FSCP-Z202)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phone-based Aftercare-Coordination (Experimental): After inpatient treatment patients receive six phone contacts of aftercare-coordination at intervals of two weeks carried out by therapists for 12 weeks. The intervention aims at supporting the patients in coordinating their aftercare treatment which can help to maintain or even improve longterm treatment outcome.
  Interventions: Behavioral: Phone-based Aftercare-Coordination
- Treatment as usual (No Intervention): After inpatient treatment patients receive treatment as usual within routine care.

INTERVENTIONS:
Behavioral: Phone-based Aftercare-Coordination — After inpatient treatment patients receive six phone contacts of aftercare-coordination at intervals of two weeks carried out by therapists for 12 weeks. The intervention is case-management orientated and aims at supporting the patients in finding and organising an adequate aftercare treatment.
  Arms: Phone-based Aftercare-Coordination

SUMMARY:
The primary objective of this study is to test in a randomized controlled trial if aftercare-coordination by phone subsequent to inpatient treatment is an effective aftercare approach in the treatment of depression and anxiety.

DETAILED DESCRIPTION:
Depression and anxiety are among the most prevalent mental health problems and are associated with a high risk of chronification. Despite the large capacities in the German health care system only a small percentage of these patients receive treatment. Relevant barriers on the pathways of patients are communication und coordination difficulties between different services and providers.The aftercare subsequent to an inpatient treatment represents one of these interfaces. Here the aim is to consolidate the treatment outcomes and to minimize the so called rebound-effect, the reduction of the positive treatment effects after the inpatient treatment. Although evidence-based treatments for depression and anxiety disorders exist, treatment effects often decrease after treatment due to the lack of an integration of different steps in care. The method of a case management-based aftercare coordination by phone could be a promising approach to overcome the interface between inpatient treatment and aftercare: case management is a patient-centered and situation-based approach which comprises systematic tracking and support of patients by a case-manager. Primary goal is to coordinate and integrate services across treatment settings. This approach can help to maintain and even improve longterm treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Depressive disorder (F32.x; F33.x; F34.1) and/or Anxiety disorder (F40.0; F40.1, F41.0; F41.1) according to ICD-10

Exclusion Criteria:

* Concurrent outpatient psychotherapeutic treatment which will be continued after the inpatient rehabilitation treatment.
* No knowledge of the German language
* Risk of suicide
* Acute psychosis or psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measure of the symptom severity - Beck Depression Inventory (BDI) | Change in the BDI from the beginning of the intervention to follow up (6 months after termination of the intervention)

SECONDARY OUTCOMES:
Measure of health related quality of life - Short Form 8 Health Survey (SF-8), Measure of health related quality of life (EQ-5D) | Change in the SF-8 and EQ-5D from the beginning of the intervention to follow up (6 months after termination of the intervention)
Proportion of patients who get routine outpatient aftercare treatment at follow up (6 months after the intervention) | 6 months after termination of the intervention
Patient-rated acceptance and satisfaction with the intervention | Approximately 3 months (end of intervention)
  Patients rate their acceptance of the intervention and their satisfaction using non-standardized items.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. phil. Hanne Melchior, Principal Investigator — University Medical Center Hamburg-Eppendorf, Centre of Psychosocial Medicine, Department of Medical Psychology
Locations (1):
- University Medical Center Hamburg-Eppendorf, Centre of Psychosocial Medicine, Department of Medical Psychology, Hamburg, Germany

REFERENCES:
- [Derived] Kivelitz L, Schulz H, Melchior H, Watzke B. Effectiveness of case management-based aftercare coordination by phone for patients with depressive and anxiety disorders: study protocol for a randomized controlled trial. BMC Psychiatry. 2015 Apr 22;15:90. doi: 10.1186/s12888-015-0469-y. PMID 25897757